CLINICAL TRIAL: NCT04360850
Title: Use of Telehealth Technology by Mental Health Care Professionals in Times of COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Hunter Hoffman, Research Scientist, Mechanical Engineering, University of Washington
Other Study IDs: STUDY00010090
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Online Therapy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: online survey — A brief survey for therapists to fill out

SUMMARY:
A brief online survey to be completed by clinical therapists.

DETAILED DESCRIPTION:
A brief online survey to be completed by clinical therapists. This brief 28 question online survey asks mental health care providers questions about their use of technology.

ELIGIBILITY:
Inclusion Criteria:

• Must be 18 years old, and must be a licensed mental healthcare provider actively treating patients within the past year.

Exclusion Criteria:

• Less than 18 years old, or if you are not a licensed mental healthcare provider actively treating patients within the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult clinical psychologists
Sampling Method: Non-Probability Sample
Enrollment: 818 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
responses to the survey questions | measured at the time they take the survey, data collection will continue for up to 1 year.
  we are not reporting an overall score on a scale, mostly true false and multiple choice

CONTACTS AND LOCATIONS:
Overall Officials: Hunter Hoffman, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sampaio M, Navarro Haro MV, Wilks C, De Sousa B, Garcia-Palacios A, Hoffman HG. Spanish-Speaking Therapists Increasingly Switch to Telepsychology During COVID-19: Networked Virtual Reality May Be Next. Telemed J E Health. 2021 Aug;27(8):919-928. doi: 10.1089/tmj.2021.0124. Epub 2021 Jun 28. PMID 34182825
- [Result] Sampaio M, Haro MVN, De Sousa B, Melo WV, Hoffman HG. Therapists Make the Switch to Telepsychology to Safely Continue Treating Their Patients During the COVID-19 Pandemic. Virtual Reality Telepsychology May Be Next. Front Virtual Real. 2021 Jan;1:576421. doi: 10.3389/frvir.2020.576421. Epub 2021 Jan 15. PMID 33585834